CLINICAL TRIAL: NCT01681342
Title: Prospective Study on the Sparing of Organs at Risk in High Dose Rate Brachytherapy for Cervix Cancer
Brief Title: Sparing of Organs at Risk in High Dose Rate Brachytherapy
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: BRACHY-HDR
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Cervical Carcinoma Stage IB to IV
Keywords: stade Ib to IV cervix cancer; ambulatory high dose rate brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cervix carcinoma is a common malignancy. Radiation therapy still remains a major treatment for patients with carcinoma cervix. Conventional treatment with radiation therapy includes a combination of external beam radiation therapy and intracavitary treatment. Low dose rate intracavitary brachytherapy treatment is already well studied. But high dose rate brachytherapy is a relatively new alternative.

In brachytherapy, major developments have been made in the integration of 3D imaging and computerized 3D treatment planning. Medical imaging improvements allowed for better definition of tumoral volumes and organs at risk.

The GYN GEC-ESTRO published recommendations on the 3D imaging for better characterization of these volumes. Improvements in CT-SCan and lately in RMN had lead to a better definition of volums of interest (tumor and his extensions and organs at risk : bladder, rectum, sigmoidis, small bowels). RMN is the imaging standard in the evaluation of tumoral extension in cervix cancer. However its use is not easy in many brachytherapy departments.

This study will evaluate the feasibility and sparing of organs at risk for high dose rate brachytherapy if volume delineation is done at each of the two sessions performed with 3D RMN.

DETAILED DESCRIPTION:
After 60 Gy are delivered with Intensity Modulated Radiation Therapy (IMRT), the brachytherapy in high dose rate will deliver 15 Gy to the CTVhr (high risk CTV) in two sessions.

A clinical examination and an RMN are performed at the end of the external radiation to evaluate the residual tumoral volume. Two HDR brachytherapy sessions are then performed.

During the first session, a CT-Scan and an RMN will be performed after the fletcher application. A second CT-Scan will be performed during the second treatment session to create new volumes and to improve organs at risk sparing.

ELIGIBILITY:
Inclusion Criteria:

* Cervix carcinoma stage Ib to IV (FIGO)
* OMS < 2
* Tomography by positron emission and/or chirurgical staging before the external radiotherapy
* RMN before the starting of treatment and at the end af external radiotherapy
* Patient information
* Validation of the indication af high dose rate brachytherapy
* External radiation therapy (60 Gy with IMRT)

Exclusion Criteria:

* No external radiation therapy
* Surgery in the 4 weeks before before the inclusion
* Prior pelvic radiation therapy
* intestinal inflammatory disease or active pathology
* active infection or severe pathology didn't allow the treatment
* Prior carcinoma in the last 5 years (except cutaneous carcinoma or in situ carcinoma)
* Inclusion in another clinical trial

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication of HDR brachytherapy in cervix carcinoma of stage IB to II.
  After realization of external radiation therapy done (60 Gy in IMRT)
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the sparing of organs at risk with a delineation at each session and the CTVhr volume modification | At 8 weeks of external radiotherapy
  To record the irradiated volumes modifications of each OAR at each session and the CTV volume modification.

SECONDARY OUTCOMES:
Evaluation of medical imaging with CT-Scan and RMN for cervix cancer | At 8 weeks of external radiotherapy
  * Interest of RMN sequences Water and T2 for the definition of volumes
  * Evaluation of imaging registration on the planning treatment system based on the brachytherapy applicator for the precision of volumes delineation
  * Evaluate the interest of TDM and RMN for volumes delineation

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Nickers, MD, PhD, Study Director — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France